CLINICAL TRIAL: NCT04212039
Title: Pericapsular Nerve Group (PENG) Block for Congenital Hip Dislocation Surgery: Randomized Controlled Double Blind Study
Brief Title: Pericapsular Nerve Group (PENG) Block for Congenital Hip Dislocation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AUTFANESTHESIAHIP
Record Dates: First submitted 2019-12-24; First posted 2019-12-26 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Congenital Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation, Congenital | interventions — Saline Solution; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided pericapsular nerve group block (Active Comparator): Ultrasound guided 0.5 ml/kg % 0.250 bupivacaine injection between to iliopubic eminentia and psoas tendon
  Interventions: Drug: Bupivacaine
- ultrasound guided sham block (Sham Comparator): Ultrasound guided 0.5 ml/kg saline injection injection between to iliopubic eminentia and psoas tendon
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Saline Solution — 0.5 ml/kg saline
  Arms: ultrasound guided sham block
Drug: Bupivacaine — 0.5 ml/kg %0.25 bupivacaine
  Arms: ultrasound guided pericapsular nerve group block

SUMMARY:
Developmental dysplasia of the hip (DDH) is one of the major disorder of the pediatric population with an incidence of 3 to 5 per 1000 children. Open surgical reduction of congenital hip dislocation (CHD) is typically performed after an ineffective closed reduction or older than 18 months. Multiple femoral or pelvic osteotomies and tenotomies are performed during this surgical treatment and cause severe postoperative pain. Pericapsular nerve group (PENG) block has been recently recommended for use as postoperative analgesia in hip surgeries. It is a new regional anesthesia method based on blocking the articular branches of femoral nerve (FN) and accessory obturator nerve (AON) in the region between the anterior inferior iliac spine (AIIS) and iliopubic eminence (IPE).The aim of this study was to evaluate the analgesic effect of ultrasound guided pediatric pericapsular nerve group (PENG) block in pediatric patients undergoing CHD surgery.

ELIGIBILITY:
Inclusion Criteria:

-American Society of Anesthesiologist's physiologic state I-II patients undergoing hip dislocation surgery

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases
* Incomplete patient forms
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* American Society of Anesthesiologist's III-IV

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry and Consolability Score (FLACC) | Postoperative first 24hour
  FLACC scale will be used. The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
Need for rescue analgesic | 2 hour
  Number of patients who required rescue analgesia in postoperative care unit in the first 2 hour
Need for analgesic | 24 hour
  Number of patients who required analgesic in the first 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aksu C, Cesur S, Kus A. Pericapsular nerve group (PENG) block for postoperative analgesia after open reduction of pediatric congenital dysplasia of the hip. J Clin Anesth. 2020 May;61:109675. doi: 10.1016/j.jclinane.2019.109675. Epub 2019 Dec 1. No abstract available. PMID 31796372
- [Background] Ahiskalioglu A, Aydin ME, Celik M, Ahiskalioglu EO, Tulgar S. Can high volume pericapsular nerve group (PENG) block act as a lumbar plexus block? J Clin Anesth. 2020 May;61:109650. doi: 10.1016/j.jclinane.2019.109650. Epub 2019 Nov 12. No abstract available. PMID 31732426
- [Background] Orozco S, Munoz D, Jaramillo S, Herrera AM. Pediatric use of Pericapsular Nerve Group (PENG) block for hip surgical procedures. J Clin Anesth. 2019 Nov;57:143-144. doi: 10.1016/j.jclinane.2019.04.010. Epub 2019 Apr 22. No abstract available. PMID 31022606
- [Background] Ahiskalioglu A, Aydin ME, Ahiskalioglu EO, Tuncer K, Celik M. Pericapsular nerve group (PENG) block for surgical anesthesia of medial thigh. J Clin Anesth. 2020 Feb;59:42-43. doi: 10.1016/j.jclinane.2019.06.021. Epub 2019 Jun 15. No abstract available. PMID 31212123
- [Background] Ahiskalioglu A, Aydin ME, Ozkaya F, Ahiskalioglu EO, Adanur S. A novel indication of Pericapsular Nerve Group (PENG) block: Prevention of adductor muscle spasm. J Clin Anesth. 2020 Mar;60:51-52. doi: 10.1016/j.jclinane.2019.08.034. Epub 2019 Aug 21. No abstract available. PMID 31445179